CLINICAL TRIAL: NCT03819426
Title: Walking or High Intensity Exercise for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01277
Record Dates: First submitted 2018-10-29; First posted 2019-01-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Social Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): Participants will be shown the appropriate techniques and intensity (high intensity; i.e., 70-90% of maximum heart rate (220-age) with a verified online youtube video. Participants will be provided with this video and other options that can be followed to complete 15 minute HIIT interventions at home. Interventionist will observe participant engaging in HIIT for 15 minutes. HIIT intervention (for 15 minutes) will also be observed during Session 4 and 8.
  Interventions: Behavioral: High Intensity Intervention
- Walking (Experimental): This intervention will be demonstrated during Session 1. Participants will be shown the appropriate walking intensity (low intensity; i.e., approximately 50% of maximum heart rate (220-age) or lower) by interventionist. Interventionist will observe participant engaging in walking at appropriate intensity level for 15 minutes. Walking intervention (for 15 minutes) will also be observed during Session 4 and 8.
  Interventions: Behavioral: Low Intensity Exercise Intervention

INTERVENTIONS:
Behavioral: Low Intensity Exercise Intervention — Those in the walking intervention will be instructed to take walks below a brisk pace (low intensity) to improve mood
  Arms: Walking
Behavioral: High Intensity Intervention — Instructed in high intensity interval training techniques and will be provided videos to follow for implementation of intervention at home that will include short bursts of high energy
  Arms: High Intensity Interval Training

SUMMARY:
After an initial phone screen process, approximately 50 participants will be enrolled and evaluated/screened in person after consenting to achieve 30 eligible participants with a principal diagnosis of GAD, panic disorder, or social anxiety disorder and high anxiety sensitivity (Anxiety Sensitivity Index score =20). Participants will be given a choice of either high intensity interval training (HIIT) or walking interventions, which will be completed over the course of 8 weeks. The goal of the study is to 1) obtain pilot data comparing the efficacy of HIIT vs. walking for effects on psychiatric, functioning and immune outcomes, 2) to identify adherence levels given the choice of exercise intensity, and 3) to identify proportion of individuals opting for each intervention. Results from this pilot study will be used to inform future grant applications including a K award.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety Sensitivity Index score of ≥20 (i.e., high anxiety sensitivity)
* Primary psychiatric diagnosis of generalized anxiety disorder (GAD), social anxiety disorder, or panic disorder
* Currently sedentary (≤60 minutes of moderate intensity exercise per week for the past 3 months)
* Able and willing to provide informed consent

Exclusion Criteria:

* Lifetime history of Bipolar I or II or any psychotic disorder
* Meets criteria for bulimia or anorexia in the past 6 months
* Meets criteria for substance use disorder in the past 3 months
* High current suicide risk as indicated by a score of ≥4 on the C-SSRS
* Risk for exercise according to Physical Activity Readiness Questionnaire with excluded medical conditions including heart conditions, lung disease, bone/joint problems, or seizures
* Women who are currently pregnant or plan to become pregnant during the duration of the study
* Participation in concurrent evidence-based therapy (e.g., cognitive behavioral therapy) targeting anxiety or depression (supportive therapy and couples therapy are allowed)
* Participants on psychiatric medication must be on a stable dose for ≥8 weeks prior to participation
* Current substance abuse or positive urine toxic screen (recreational use of marijuana is permitted based on clinical assessment on the MINI that it does not meet criteria for cannabis use disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of HIIT measured by Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q-SF) | Week 1
  Scoring involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are stand alone items. The raw score ranges from 14 to 70.
Efficacy of HIIT measured by Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q-SF) | Week 10
  Scoring involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are stand alone items. The raw score ranges from 14 to 70.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Szuhany, PhD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Any requests for data will be considered on a case by case basis given the pilot nature of this project. As this is a pilot study, there will not be sufficient data for systematic sharing. Means of participant data will be shared on clinicaltrials.gov.
Time Frame: On a case by case basis, given the pilot nature of this project.
Access Criteria: Requests should be directed to Kristin.szuhany@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.